CLINICAL TRIAL: NCT04498676
Title: 50 Human Subject Repeat Insult Patch Test Skin Irritation/Sensitization Evaluation (Occlusive Patch)
Brief Title: 50 Human Subject Repeat Insult Patch Test
Acronym: HRIPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CAGE Bio Inc. (Industry)
Collaborators: AMA Laboratories Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: MS17.RIPT.P1200O.50.CBIO
Record Dates: First submitted 2020-07-29; First posted 2020-08-04 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-07

CONDITIONS: Erythema; Sensitisation
Keywords: HRIPT; irritant
MeSH Terms: conditions — Erythema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Test product (Experimental)
  Interventions: Other: CB-0002B

INTERVENTIONS:
Other: CB-0002B — CB-0002B (choline geranate) is a viscous transparent colorless to light yellow liquid

SUMMARY:
Consumer products or raw materials designed for consistent reapplication to areas of the skin may, under proper conditions, prove to be contact sensitizers or irritants in certain individuals. It is the intention of a Repeat Insult Patch Test (RIPT) to provide a basis for evaluation of this irritation/sensitization potential if such exists.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who are not currently under a doctor's care
* Individuals free of any dermatological or systemic disorder which would interfere with the results, at the discretion of the Investigator.
* Individuals free of any acute or chronic disease that might interfere with or increase the risk of study participation.
* Individuals who will complete a preliminary medical history form mandated by AMA Laboratories, Inc. and are in general good health.
* Individuals, who will read, understand and sign an informed consent document relating to the specific type of study they are subscribing. Consent forms are kept on file and are available for examination on the premises of AMA Laboratories, Inc. only.
* Individuals able to cooperate with the Investigator and research staff, willing to have test materials applied according to the protocol, and complete the full course of the study.

Exclusion Criteria:

* Individuals under 18 years of age.
* Individuals who are currently under a doctor's care.
* Individuals who are currently taking any medication (topical or systemic) that may mask or interfere with the test results.
* Subjects with a history of any acute or chronic disease that might interfere with or increase the risk associated with study participation.
* Individuals diagnosed with chronic skin allergies.
* Female volunteers who indicate that they are pregnant or lactating.

Ages: 21 Years to 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-01-18 (Actual); Primary Completion 2017-02-08 (Actual); Study Completion 2017-03-02 (Actual)

PRIMARY OUTCOMES:
Erythema | 21 days
  Erythema rated on a numeric scale from 0 - 4. (0: None; 1: Minimal; 2: Mild; 3: Marked and 4: Severe erythema)
Sensitisation | 24 hours
  After a 10-14 day rest period, a challenge test was given at a different skin site to look for signals of a sensitization response measured by rating erythema on a scale from 0 - 4
Sensitisation | 48 hours
  After a 10-14 day rest period, a challenge test was given at a different skin site to look for signals of a sensitization response measured by rating erythema on a scale from 0 - 4

CONTACTS AND LOCATIONS:
Overall Officials: Director, Study Director — AMA Laboratories Inc.
Locations (1):
- AMA Laboratories Inc., New City, New York, United States

IPD SHARING:
Plan to Share IPD: No